CLINICAL TRIAL: NCT07124910
Title: Comparison of Epi-ON Corneal Collagen Crosslinking Performed Using an 18-Minute UVA Exposure Versus a 24-Minute UVA Exposure on Eyes With Ectatic Corneal Diseases
Brief Title: Comparison of Epi-ON Corneal Collagen Crosslinking Performed Using an 18-Minute UVA Exposure vs. a 24-Minute UVA Exposure on Eyes With Ectatic Corneal Diseases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Woolfson Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WEI-CXL-003
Record Dates: First submitted 2025-08-05; First posted 2025-08-15 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Keratoconus; Ectasia of Cornea; Pellucid Marginal Corneal Degeneration; Forme Fruste Keratoconus (FFK)
Keywords: crosslinking; corneal; Epi-ON; UVA
MeSH Terms: conditions — Keratoconus | interventions — Corneal Cross-Linking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- UVA 18 minute (Experimental): Subjects who meet the inclusion criteria and provide informed consent will be randomized to receive UVA irradiation with 15-second off-on cycling for either 18 minutes or 24 minutes
  Interventions: Combination Product: Epi-ON corneal cross-linking
- UVA 24 minute (Experimental): Subjects who meet the inclusion criteria and provide informed consent will be randomized to receive UVA irradiation with 15-second off-on cycling for either 18 minutes or 24 minutes
  Interventions: Combination Product: Epi-ON corneal cross-linking

INTERVENTIONS:
Combination Product: Epi-ON corneal cross-linking — Corneal cross-linking involves the following steps:
  * applying riboflavin (Vitamin B2 eye drops) to the eye, then
  * exposing the eye to ultraviolet (UV-A) light

SUMMARY:
The goal of this clinical trial is to study the effects of an experimental (not Food and Drug Administration (FDA)-approved) treatment called corneal crosslinking (CXL) for conditions in which the cornea becomes progressively thin, steep, and misshapen, causing vision to be blurred.

CXL is performed by putting riboflavin (vitamin B2) drops onto the eye and then exposing it to ultraviolet (UVA) light at about the same intensity as you get outdoors on a bright, sunny day. It is designed to stop the progression of disease by strengthening the cornea. Study participants will be at least 8 years of age or older and have a diagnosis of keratoconus, ectasia after LASIK, ectasia after PRK, pellucid marginal degeneration, progressive ectasia after previous CXL treatment or forme fruste keratoconus.

The main question it aims to answer is:

* Does CXL help prevent or slow the progression of someone's corneal condition and vision loss?

Participants will:

* Attend up to a total of 7 in office visits over the course of 6 months, where several eye and vision tests will be given.

Receive CXL (applying riboflavin (Vitamin B2 eye drops) to the eye, then exposing the eye to ultraviolet (UV-A) light).

* There will be two groups of participants. One group will receive the UVA treatment for 18 minutes and the other group will receive the UVA treatment for 24 minutes.

ELIGIBILITY:
Inclusion Criteria:

Subjects in whom both the subject and study eye meet all of the following criteria are candidates for the study:

1. Be at least 8 years of age or older, male or female, of any race.
2. Have a diagnosis of keratoconus, ectasia after LASIK, ectasia after PRK, pellucid marginal degeneration, progressive ectasia after previous CXL treatment or forme fruste keratoconus based on topography, tomography, and slit lamp examination.
3. Provide written informed consent and a signed HIPAA form. Pediatric subjects less than 14 years of age must sign an assent, and a parent or legal guardian must sign an informed consent.
4. Be willing and able to follow all instructions and comply with the schedule for follow-up visits.
5. If female and capable of becoming pregnant, must not be lactating or pregnant and must agree to use a medically acceptable form of birth control for at least one week prior to the treatment visit and to continue one month following treatment.

Exclusion Criteria:

Subjects in whom the subject or study eye meets one or more of the following criteria will be excluded from the randomized cohort of the study:

1. Normal corneal topography.
2. A history of previous corneal transplant in the study eye.
3. Minimum corneal thickness < 300 (measured by Pentacam and Ultrasound) at the screening exam.
4. Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye to future complications or prevent the possibility of improved vision, for example:

   1. History of or active corneal disease (e.g., herpes simplex, herpes zoster keratitis, etc.)
   2. Clinically significant corneal scarring in the central cornea that, in the investigator's opinion, will not allow the subject to achieve functional vision, even with contact lens correction, after the crosslinking procedure.
5. A known contraindication, sensitivity, or allergy to the test article or its components or to study medications.
6. Nystagmus or any other condition that would prevent a steady gaze during the crosslinking treatment or other diagnostic tests.
7. If female, pregnant, nursing or planning a pregnancy, or having a positive urine pregnancy test prior to the randomization of, or treatment of either eye during the course of the study.
8. Inability to remove soft or scleral contact lenses at least 3 days before initial and follow-up examinations.
9. Inability to remove rigid gas-permeable contact lenses at least 2 weeks before initial and follow-up examinations.
10. Inability to return for required postoperative examinations.
11. Presence or history or any other condition or finding that, in the investigator's opinion, makes the subject unsuitable as a candidate for crosslinking or study participation or may confound the outcome of the study.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 485 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary outcome measures for efficacy is corneal curvature, as measured by Kmax with the Pentacam, in the treated eyes and CDVA. | From enrollment to the end of treatment at 6 months.
  The change in keratometry (Kmax) and corrected visual acuity from baseline will be evaluated at 6 months for all eyes treated. Data will be summarized using descriptive statistics and experimental groups will be compared using nonparametric tests. The change in Kmax and corrected visual acuity from baseline will be evaluated at 6 months.

SECONDARY OUTCOMES:
Change in UCVA compared to the baseline examination will be used as a Secondary outcome measurement. | 6 months
  Change in UCVA compared to the baseline examination will be evaluated at 6 months postoperatively. Data will be summarized using descriptive statistics and experimental groups will be compared using nonparametric tests.
At the Sponsor-Investigator's discretion, the change in HOA from baseline may be evaluated at 6 months postoperatively for the eyes that underwent preoperative and postoperative wavefront testing. | 6 months
  Data will be summarized using descriptive statistics and experimental groups will be compared using nonparametric tests.
At the Sponsor-Investigator's discretion, the change in coma from baseline may be evaluated at 6 months postoperatively for the eyes that underwent preoperative and postoperative wavefront testing. | 6 months
  Data will be summarized using descriptive statistics and experimental groups will be compared using nonparametric tests.

CONTACTS AND LOCATIONS:
Locations (11):
- United States (11):
  - Woolfson Eye Institute, Atlanta, Georgia
  - Woolfson Eye Institute, Canton, Georgia
  - Woolfson Eye Institute, Cumming, Georgia
  - Woolfson Eye Institute, Douglasville, Georgia
  - Woolfson Eye Institute, Lawrenceville, Georgia
  - Woolfson Eye Institute, Marietta, Georgia
  - Woolfson Eye Institute, Snellville, Georgia
  - Woolfson Eye Institute, Asheville, North Carolina
  - Woolfson Eye Institute, Chattanooga, Tennessee
  - Woolfson Eye Institute, Johnson City, Tennessee
  - Woolfson Eye Institute, Knoxville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided